CLINICAL TRIAL: NCT00688753
Title: A Single Arm, Multicenter Phase II Trial of RAD001 as Monotherapy in the Treatment of Advanced Papillary Renal Cell Cancer
Brief Title: RAPTOR: RAD001 as Monotherapy in the Treatment of Advanced Papillary Renal Cell Tumors Program in Europe
Acronym: MACS0460
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001LFR08; 2008-006181-28
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma; Renal Cell; Non Clear Cell Renal Carcinoma; Papillary Cell Renal Carcinoma; Adenocarcinoma
Keywords: renal cell carcinoma; non clear cell carcinoma; papillary cell renal carcinoma; adults; everolimus
MeSH Terms: conditions — Carcinoma; Carcinoma, Renal Cell; Adenocarcinoma | interventions — Everolimus

ARMS (1):
- RAD001 (Experimental): two 5 mg tablets of everolimus orally, once daily
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001

SUMMARY:
To evaluate the preliminary efficacy and safety of RAD001 as monotherapy for first-line treatment of patients with metastatic papillary carcinoma of the kidney.

ELIGIBILITY:
Inclusion criteria:

1. ≥ 18 years old.
2. Patients with metastatic papillary renal cell carcinoma, type I or II.
3. Patients with at least one measurable lesion.
4. Patients with an ECOG Performance Status ≤1.
5. Adequate bone marrow function.
6. Adequate liver function.
7. Adequate renal function.
8. Adequate lipid profile.

Exclusion criteria:

1. Patients who had radiation therapy within 28 days prior to start of study.
2. Patients who have received prior systemic treatment for their metastatic RCC.
3. Patients who received prior therapy with VEGF pathway inhibitor.
4. Patients who have previously received systemic mTOR inhibitors.
5. Patients with a known hypersensitivity everolimus or other rapamycins or to its excipients.
6. Patients with uncontrolled central nervous system (CNS) metastases.
7. Patients receiving chronic systemic treatment with corticosteroids or another immunosuppressive agent.
8. Patients with a known history of HIV seropositivity.
9. Patients with autoimmune hepatitis.
10. Patients with an active, bleeding diathesis.
11. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
12. Patients who have a history of another primary malignancy and off treatment ≤ 3 years, with the exception of non-melanoma skin cancer and carcinoma in situ of the uterine cervix.
13. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
14. Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to study treatment start.
15. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Münster
- Italy (4):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Otwock, Poland
- Spain (3):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

REFERENCES:
- [Derived] Escudier B, Molinie V, Bracarda S, Maroto P, Szczylik C, Nathan P, Negrier S, Weiss C, Porta C, Grunwald V, Albiges L. Open-label phase 2 trial of first-line everolimus monotherapy in patients with papillary metastatic renal cell carcinoma: RAPTOR final analysis. Eur J Cancer. 2016 Dec;69:226-235. doi: 10.1016/j.ejca.2016.08.004. Epub 2016 Sep 24. PMID 27680407

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: two 5 mg tablets orally, once daily at the same time every day immediately after a meal
Period: Overall Study
Arm/Group | RAD001
Started | 92
Completed | 0
Not Completed | 92
Not completed — Disease progression | 55
Not completed — Missing | 1
Not completed — Death | 9
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 20
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- RAD001 10 mg: two 5 mg tablets of everolimus orally, once daily
Arm/Group | RAD001 10 mg
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Efficacy of RAD001 as Monotherapy for the Treatment of Papillary Renal Cancer. Efficacy is Defined as the Percentage of Patients Progression-free at 6 Months.
Description: PFSR at 6 months based on central review
Time Frame: 6 mos
Population: PP, PPFF, ITT
Measure: Number (80% Confidence Interval); unit: % participants
Groups:
- RAD001: 10 mg/day
Arm/Group | RAD001
Number analyzed (Participants) | 92
% participants
  (PPFF Set, N=44) | 34.1 [24.5 to 44.8]
  (PPSet, N=66) | 33.3 [25.6 to 41.8]
  (ITT Set, N=86) | 32.6 [25.9 to 39.9]

2. Secondary Outcome: Disease Control Rate (SD + PR + CR)
Description: DCR was defined as the proportion of patients with a best overall response of CR, PR or SD and ORR as the percentage of patients with CR or PR
Time Frame: 6 mos
Population: PP,ITT
Measure: Number (90% Confidence Interval); unit: % Participants
Arm/Group | RAD001
Number analyzed (Participants) | 92
% Participants
  PP set | 65.2 [54.4 to 74.9]
  ITT set | 65.1 [55.8 to 73.6]

3. Secondary Outcome: Objective Response Rate
Description: ORR is defined as the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period. Response duration usually is measured from the time of initial response until documented tumor progression
Time Frame: End of trial
Measure: Number (90% Confidence Interval); unit: % participants
Arm/Group | RAD001
Number analyzed (Participants) | 92
% participants
  PP Set | 1.5 [0.1 to 7.0]
  ITT Set | 1.2 [0.1 to 5.4]

4. Secondary Outcome: Duration of Response
Description: The DOR analysis applied only to patients whose overall response was CR or PR and was defined as the time from onset of response (CR/PR) to progression or death from any cause.
Time Frame: End of trial
Population: In the final analysis, for central review, the DOR could not be calculated as only 1 patient in the PP and ITT sets met the criteria
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RAD001
Number analyzed (Participants) | 92
days
  local review PP set | 169 [64 to 169]
  local review ITT set | 226 [64 to 928]

5. Secondary Outcome: Median Progression Free Survival
Description: PFS was defined as the time from first study drug administration to objective tumor progression or death from any cause.
Time Frame: End of trial
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RAD001
Number analyzed (Participants) | 92
days
  PP set | 118 [65 to 174]
  ITT set | 113 [77 to 167]

6. Secondary Outcome: Incidence of Adverse Events, Serious Adverse Events, and Death.
Time Frame: End of trial
Population: Safety Set
Measure: Number; unit: % participants
Arm/Group | RAD001
Number analyzed (Participants) | 92
% participants
  Patients with any AE | 100
  AE with suspected relation to study drug | 97.83
  AE leading to dose adjustment or interruption | 53.26
  AE leading to permanent discontinuation | 27.17
  AE requiring concomitant medication | 90.22
  Patients with serious adverse event (SAE) | 46.74
  SAE suspected relation to study drug | 23.91
  SAE leading to permanent discontinuation | 10.87
  Patients died | 10.87

ADVERSE EVENTS:
Groups:
- All Patients: two 5 mg tablets orally, once daily at the same time every day immediately after a meal
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 43/92
Other Adverse Events (participants affected / at risk) | 90/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=92)
Anaemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 4
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 2
General physical health deterioration (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 4
Cholestasis (Hepatobiliary disorders) | 1
Anal infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 1
Postoperative abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Aphasia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Renal failure acute (Renal and urinary disorders) | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=92)
Anaemia (Blood and lymphatic system disorders) | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Tachycardia (Cardiac disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 23
Aphthous stomatitis (Gastrointestinal disorders) | 11
Ascites (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 36
Dry mouth (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 27
Stomatitis (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 39
Chest pain (General disorders) | 7
Fatigue (General disorders) | 30
Mucosal inflammation (General disorders) | 36
Oedema peripheral (General disorders) | 29
Pain (General disorders) | 7
Pyrexia (General disorders) | 25
Bronchitis (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood creatinine increased (Investigations) | 8
Platelet count decreased (Investigations) | 6
Weight decreased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 36
Hypercholesterolaemia (Metabolism and nutrition disorders) | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 12
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dysgeusia (Nervous system disorders) | 23
Headache (Nervous system disorders) | 16
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 12
Nail disorder (Skin and subcutaneous tissue disorders) | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 53
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.